CLINICAL TRIAL: NCT02039180
Title: A Phase 1, Open-label, Randomized, Single-dose, 3-period Cross-over, Relative Bioavailability Study to Assess Two Solid Formulations Compared to an Oral Solution of AZD3293 in Healthy Male and Non-Fertile Female Subjects
Brief Title: Relative Bioavailability Study to Assess Two Solid Formulations Compared to an Oral Solution of AZD3293 in Healthy Male and Non-Fertile Female Subjects
Acronym: BA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5010C00005
Record Dates: First submitted 2014-01-16; First posted 2014-01-17 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers; Pharmacologic Action
Keywords: phase I; healthy volunteers; AZD3293; bioavailability; Pharmacokinetics
MeSH Terms: interventions — lanabecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD3293 oral solution (Experimental): single doses in random order in 3 study periods for each subject (Day 1 or Day 8 or Day 15)
  Interventions: Drug: AZD3293 oral solution
- AZD3293 tablet formulation A (Experimental): single doses in random order in 3 study periods for each subject (Day 1 or Day 8 or Day 15)
  Interventions: Drug: AZD3293 tablet formulation A
- AZD3293 tablet formulation B (Experimental): single doses in random order in 3 study periods for each subject (Day 1 or Day 8 or Day 15)
  Interventions: Drug: AZD3293 tablet formulation B

INTERVENTIONS:
Drug: AZD3293 oral solution — Subjects will receive AZD3293 as a tablet (Formulation A; Formulation B) and solution as a single dose on Day 1, Day 8 or Day 15.
  Other Names: Beta secretase inhibitor
  Arms: AZD3293 oral solution
Drug: AZD3293 tablet formulation A — Subjects will receive AZD3293 as a tablet (Formulation A; Formulation B) and a solution as a single dose on Day 1, Day 8, or Day 15.
  Other Names: beta secretase inhibitor
  Arms: AZD3293 tablet formulation A
Drug: AZD3293 tablet formulation B — Subjects will receive AZD3293 as a tablet (Formulation A; Formulation B) and a solution as a single dose on Day 1, Day 8 or Day 15.
  Other Names: Beta secretase inhibitor
  Arms: AZD3293 tablet formulation B

SUMMARY:
This is an open-label, randomized, 3-period crossover, single dose study. Three (3) single doses of AZD3293 (2 different tablet formulations, and an oral solution) will be administered with a washout period of at least 1 week between the doses to investigate the relative bioavailability of AZD3293 after administration via 2 tablet formulations compared with oral solution and to evaluate basic systemic pharmacokinetic parameters of the tablet formulations compared to the oral solution of AZD3293.

The safety and tolerability of AZD3293 in healthy subjects will also be assessed in the study. AZD3293 is being developed for the treatment of Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written, and dated informed consent prior to any study-specific procedures
2. Healthy subjects must be able to understand and be willing to comply with study procedures, restrictions, and requirements.
3. Male and non-fertile female healthy subjects, aged 18 to 55 years
4. Body weight ≥50 to ≤100 kg and body mass index (BMI) ≥19 to ≤30 kg/m2
5. Clinically normal findings on physical examination in relation to age, as judged by the Investigator

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
3. History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder according to the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV), as assessed by the Mini-International Neuropsychiatric Interview (MINI)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The relative bioavailability of AZD3293 after administration via 2 tablet formulations compared with oral solution by assessment of the area under the plasma concentration-time curve from zero to infinity for the tablet formulations and the oral solutio | up to day 18 (Day 1 - 72 hrs post-dose on Day 15)
  Blood samples for determination of plasma concentrations of AZD3293 and its active metabolite will be collected at pre-dose (15 or 30 min) and 30 min, 1h, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56 and 72 hours post-dose starting on Days 1, 8 & 15 and analyzed according to fully validated methods.
To compare the tablet formulations of AZD3293 with the oral solution of AZD3293 by evaluation of the basic pharmacokinetic parameters for each formulation | up to day 18 (Day 1 - 72 hrs post-dose on Day 15)
  Blood samples for determination of plasma concentrations of AZD3293 and its active metabolite will be collected at pre-dose (15 or 30 min) and 30 min, 1h, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 56 and 72 hours post-dose starting on Days 1, 8 & 15 and analyzed according to fully validated methods.

SECONDARY OUTCOMES:
Safety profile in terms of Adverse events assessment | From Baseline and up to day 25
Safety and tolerability in terms of lab tests assessment (hematology, chemistry, urinalysis) | From Baseline and up to day 25
Safety and tolerability in terms of vital signs assessment (blood pressure, pulse and body temperature) and physical exams | From baseline and up to day 25
Safety and tolerability by assessing changes in electrocardiogram (ECG) parameters | from baseline and up until day 25

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Cypress, California, United States